CLINICAL TRIAL: NCT06645483
Title: How Does ChatGPT Contribute to Improving University Students' Psychological Preparedness for Natural Disasters and Perceived Disaster Risk?: a Randomized Controlled Trial
Brief Title: ChatGPT Contribute to the Development of Psychological Preparedness and Disaster Risk Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lütfiye Parlak (Other)
Responsible Party: Sponsor-Investigator, Lütfiye Parlak, Lecturer, Kutahya Health Sciences University
Organization: Kutahya Health Sciences University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KutahyaHSU-PARLAK-043
Record Dates: First submitted 2024-09-20; First posted 2024-10-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: University Student
Keywords: disaster; risk perception; university students; chatgpt

STUDY DESIGN:
Intervention Model Description: Branch A and Branch B will be randomly assigned as the experimental and control groups via a draw conducted through the randomizer.org website. At the beginning of the study, a pre-test will be administered to both groups. The lessons for the experimental group will be conducted using ChatGPT during the first two weeks, while the control group will receive instruction through the traditional teaching method (presentation-based instruction). At the end of the two weeks, a post-test will be administered to both groups. To ensure that the students receive the same course under the same conditions and opportunities, the teaching methods will be crossed between the groups during the following two weeks, with the experimental group receiving traditional education and the control group being taught with ChatGPT. At the end of the total four-week implementation, a follow-up test will be administered to both groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ChatGPT Group (Experimental): In this group, students will receive ChatGPT-assisted education for the first two weeks of the "Emergency and Disaster Management" course. ChatGPT will be integrated into the course to answer student questions, explain topics, and provide customized content aligned with the learning objectives. For the following two weeks, students will be taught using traditional instructional methods (lecture-based teaching).
  Interventions: Other: ChatGPT-assisted instruction
- Traditional Teaching Group (Active Comparator): In this group, students will receive traditional lecture-based instruction for the first two weeks of the course. For the following two weeks, they will switch to ChatGPT-assisted education.
  Interventions: Other: Traditional lecture-based instruction

INTERVENTIONS:
Other: ChatGPT-assisted instruction — ChatGPT will interactively support students by answering questions, initiating discussions, and providing customized learning materials in line with the course objectives. It will be supervised by the instructor to ensure guidance and prevent misinformation.
  Duration: ChatGPT-assisted learning for the first two weeks, followed by traditional teaching for the next two weeks.
  Arms: ChatGPT Group
Other: Traditional lecture-based instruction — Students will learn through a traditional teaching format, where the instructor delivers the course content through lectures and presentations.
  Duration: Traditional teaching for the first two weeks, followed by ChatGPT-assisted learning for the next two weeks.
  Arms: Traditional Teaching Group

SUMMARY:
The study aims to contribute to the design of new approaches in enhancing disaster risk perception and the improvement of intervention strategies in this field by identifying the different levels of psychological preparedness among individuals.

Type, Location, and Time of the Study

This study is a randomized controlled trial that will be conducted prospectively in a cross-sectional design. It will take place at Kütahya Health Sciences University, Simav Vocational School of Health Services, during the Fall semester of the 2024-2025 academic year, involving students enrolled in the "Emergency and Disaster Management" courses.

Population and Sample The population of this study will consist of second-year students enrolled in the Fall semester of the 2024-2025 academic year at Kütahya University of Health Sciences, Simav Vocational School of Health Services (https://oidb.ksbu.edu.tr/index/sayfa/10106/ocak-2024). The "Emergency and Disaster Management" course is offered as an elective for all second-year students across the departments of Simav Vocational School of Health Services. The course is taught in two separate sections (Sections A and B) by Lecturer Dr. Nahsan KAYA.

The sample size of the study, based on the power analysis conducted using the G*Power software, will consist of 72 students, with 36 students in each group, assuming 80% power, a 0.05 margin of error, and a 1:1 randomization ratio.

Branch A and Branch B will be randomly assigned as the experimental and control groups via a draw conducted through the randomizer.org website. At the beginning of the study, a pre-test will be administered to both groups. The lessons for the experimental group will be conducted using ChatGPT during the first two weeks, while the control group will receive instruction through the traditional teaching method (presentation-based instruction). At the end of the two weeks, a post-test will be administered to both groups. To ensure that the students receive the same course under the same conditions and opportunities, the teaching methods will be crossed between the groups during the following two weeks, with the experimental group receiving traditional education and the control group being taught with ChatGPT. At the end of the total four-week implementation, a follow-up test will be administered to both groups.

DETAILED DESCRIPTION:
H1. The psychological preparedness levels of university students in the experimental group for natural disasters will be higher in the assessment conducted in the second week compared to the baseline assessment.

H1. The psychological preparedness levels of university students in the experimental group for natural disasters will be higher in the second-week assessment compared to the students in the control group.

H1. The psychological preparedness levels of university students in the control group for natural disasters will be higher in the assessment conducted in the fourth week compared to the baseline and second-week assessments.

H1. The disaster risk perceptions of university students in the experimental group will be higher in the assessment conducted in the second week compared to the baseline assessment.

H1. The disaster risk perceptions of university students in the experimental group will be higher in the second-week assessment compared to the students in the control group.

H1. The disaster risk perceptions of university students in the control group will be higher in the assessment conducted in the fourth week compared to the baseline and second-week assessments.

Data Collection Tools

Socio-demographic Characteristics and Introduction Information Form: It consists of a total of 12 questions prepared by the researchers in line with the purposes of the study. Questions 10, 11 and 12 will be answered by students using ChatCPT under the guidance of an instructor in the "Emergency and Disaster Management" course.

Psychological Preparedness for Disaster Threat Scale: The Turkish validity and reliability study of the scale developed by Zulch (2019) regarding psychological preparedness for disasters in Northern Australian communities was conducted by Türkdoğan-Görgün, Koçak-Şen and McLennan (2023). The scale consists of a total of 21 items under 3 sub-dimensions: "External Situational Environment Knowledge and Management", "Management of the Person's Emotional and Psychological Response" and "Management of the Person's Social Environment". Each item in the scale is evaluated with a 4-point Likert-type rating as 1- Strongly Disagree, 4- Strongly Agree. A minimum of 21 and a maximum of 84 points can be obtained from the scale. The Cronbach Alpha coefficient for the sub-dimensions and the overall scale are 0.91, 0.93, 0.83 and 0.95, respectively (Türkdoğan-Görgün, Koçak-Şen & McLennan, 2023).

University Students Disaster Risk Perception Scale: Developed by Mızrak and Aslan (2020) to assess the disaster risk perception of university students. The scale consists of 19 items in total under 4 sub-dimensions named "Exposure", "Anxiety", "Impact" and "Unmanageability". Each item in the scale is evaluated with a 5-point Likert-type rating as 1- Strongly Disagree and 5- Strongly Agree. A minimum of 19 and a maximum of 95 points can be obtained from the scale. Cronbach Alpha reliability coefficients for the sub-dimensions of the scale are 0.89, 0.89, 0.88 and 0.78, respectively. (Mızrak & Aslan, 2020).

Mızrak, S., & Aslan, R. (2020). Disaster risk perception of university students. Risk, Hazards & Crisis in Public Policy, 11(4), 411-433. https://doi.org/10.1002/rhc3.12202

Türkdoğan-Görgün, C., Koçak-Şen, İ., & McLennan, J. (2023). The validity and reliability of the Turkish version of the Psychological Preparedness for Disaster Threat Scale. Nat Hazards. https://doi.org/10.1007/s11069-023-06006-w

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Take an emergency disaster management course
* Volunteer to participate in the study

Exclusion Criteria:

* Refusing to participate in the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Psychological Preparedness for Disaster Threats Scale (PPDTS) - Total Score | Week 0 (at the beginning of the study), week 2, and week 4 (at the end of the study)
  Psychological Preparedness for Disaster Threats Scale (PPDTS): This scale assesses psychological preparedness for disaster threats in three subdimensions: "External Situational Awareness and Management," "Management of Emotional and Psychological Response," and "Management of Social Environment." Scores range from 21 to 84, with higher scores indicating higher levels of psychological preparedness. Data will be summarized using the total scale score as well as subdimension scores. Total score from the PPDTS, ranging from 21 to 84. This scale measures psychological preparedness across three subdimensions. The total score will be used as the primary outcome measure for preparedness.
Perceived Disaster Risk Scale for University Students (PDRSUS) - Total Score | Week 0 (at the beginning of the study), week 2, and week 4 (at the end of the study)
  Perceived Disaster Risk Scale for University Students (PDRSUS): This scale evaluates perceived disaster risk among university students across four subdimensions: "Exposure," "Anxiety," "Impact," and "Unmanageability." Scores range from 19 to 95, with higher scores indicating greater perceived risk. Data will be summarized using the total scale score and subdimension scores. Total score from the PDRSUS, ranging from 19 to 95. This scale measures perceived disaster risk across four subdimensions. The total score will be used as the primary outcome measure for risk perception

SECONDARY OUTCOMES:
Subdimension Scores on the Psychological Preparedness for Disaster Threats Scale (PPDTS) | Week 0 (at the beginning of the study), week 2, and week 4 (at the end of the study)
  Subdimension scores for "External Situational Awareness and Management," "Management of Emotional and Psychological Response," and "Management of Social Environment." Scores for each subdimension range from 3 to 12 or 9 to 36. These scores will be analyzed separately as secondary outcome measures.
Subdimension Scores on the Perceived Disaster Risk Scale for University Students (PDRSUS) | Week 0 (at the beginning of the study), week 2, and week 4 (at the end of the study)
  Subdimension scores for "Exposure," "Anxiety," "Impact," and "Unmanageability." Scores for each subdimension range from 5 to 25 or 6 to 30. These scores will be analyzed separately as secondary outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: PINAR DURU, Assoc. Prof., Study Director — pduru@ogu.edu.tr
Locations (1):
- Kütahya Health Science University, Simav Health Services Vocational School, Kütahya, Simav, Turkey (Türkiye)